CLINICAL TRIAL: NCT04675268
Title: Variability in Nocturnal Oxygen Parameters in Suspected Obstructive Sleep Apnea
Brief Title: Variability in Nocturnal Oxygen Parameters in Suspected Obstructive Sleep Apnea (OSA)
Acronym: VARIOUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s64296
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: oximetry
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7 night home oximetry (Experimental): Patients will undergo 7 nights home monitoring with oximetry.
  Interventions: Diagnostic Test: oximetry

INTERVENTIONS:
Diagnostic Test: oximetry — A CE medical approved polygraphy device (Dreamscan 2 - Medatec) will be used to obtain oximetry (and PPG) data

SUMMARY:
The investigators would like to evaluate the variability of oxygen (and PPG) parameters during 7 nights at home. Oxygen (and PPG) parameters will also be evaluated during 1 night at the hospital (diagnostic polysomnography).

Based on currently developed algorithms, surrogate apnea-hypopnea index (AHI), cardiovascular status and the variability of these parameters will be evaluated.

DETAILED DESCRIPTION:
The main objective of this trial is to evaluate the variability in nocturnal oxygen (and PPG) parameters during 7 consecutive nights at home and to identify clinical predictors of variability in patients with suspected OSA.

Data regarding sleep position, alcohol intake and sleep duration will be evaluated (these parameters could be important to explain variability).

Additional objectives are to compare the parameters measured at home with the parameters measured during an in-hospital polysomnography.

The investigators will also evaluate variability in the surrogate AHI described by the group based on the measurements at home and the impact of multi-night evaluation of oxygen (and PPG) parameters on the recently developed mICS algorithm will be explored.

This study is a first explorative approach for further (multi-site) work to define the burden of OSA associated with cardiovascular or psychofunctional problems.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected OSA with a clinical indication to perform a polysomnography

Exclusion Criteria:

* Patients younger than 18 yrs
* Patients not able to read or understand the informed consent content on the purpose of the study, due to visual, intellectual or language issues
* Patients with neuromuscular disease or chest wall disease with suspected hypoventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Variability in oxygen desaturation index 3 percent | 7 nights
  Using a CE medical approved polygraphy device (Dreamscan 2 - Medatec) the variability in number of oxygen desaturation events with desaturation higher or equal to 3% is evaluated.
  Mean +/- SD or median (interquartile range) depending whether or not the 7 night data present a Gaussian distribution, and the coefficient of variation (CV).
Variability in oxygen desaturation index 4 percent | 7 nights
  Using a CE medical approved polygraphy device (Dreamscan 2 - Medatec) the variability in number of oxygen desaturation events with desaturation higher or equal to 4% is evaluated.
  Mean +/- SD or median (interquartile range) depending whether or not the 7 night data present a Gaussian distribution, and the coefficient of variation (CV).
Variability in mean oxygen saturation | 7 nights
  Using a CE medical approved polygraphy device (Dreamscan 2 - Medatec) the variability in mean nocturnal oxygen saturation during 7 consecutive nights at home is evaluated.
  Mean +/- SD or median (interquartile range) depending whether or not the 7 night data present a Gaussian distribution, and the coefficient of variation (CV).
Variability in minimal oxygen saturation | 7 nights
  Using a CE medical approved polygraphy device (Dreamscan 2 - Medatec) the variability in mean nocturnal oxygen saturation during 7 consecutive nights at home is evaluated.
  Mean +/- SD or median (interquartile range) depending whether or not the 7 night data present a Gaussian distribution, and the coefficient of variation (CV).
Variability in percentage of time oxygen saturation < 90 percent | 7 nights
  Using a CE medical approved polygraphy device (Dreamscan 2 - Medatec) the variability in mean nocturnal oxygen saturation during 7 consecutive nights at home is evaluated.
  Mean +/- SD or median (interquartile range) depending whether or not the 7 night data present a Gaussian distribution, and the coefficient of variation (CV).
Variability in percentage of time oxygen saturation < 88 percent | 7 nights
  Using a CE medical approved polygraphy device (Dreamscan 2 - Medatec) the variability in mean nocturnal oxygen saturation during 7 consecutive nights at home is evaluated.
  Mean +/- SD or median (interquartile range) depending whether or not the 7 night data present a Gaussian distribution, and the coefficient of variation (CV).
Variability in percentage of time oxygen saturation < 80 percent | 7 nights
  Using a CE medical approved polygraphy device (Dreamscan 2 - Medatec) the variability in mean nocturnal oxygen saturation during 7 consecutive nights at home is evaluated.
  Mean +/- SD or median (interquartile range) depending whether or not the 7 night data present a Gaussian distribution, and the coefficient of variation (CV).

SECONDARY OUTCOMES:
Evaluation of clinical predictors (alcohol intake, sleep duration) of this variability. | 7 nights
  Based on sleep diaries, the correlation between alcohol intake and/or sleep duration and the variability of nocturnal oxygen parameters is evaluated.
Evaluation of clinical predictors (body position) of this variability. | 7 nights
  Based on data of the McRoberts Move monitor, the correlation between body position and the variability of nocturnal oxygen parameters is evaluated.
To compare nocturnal oxygen (and PPG) parameters measured at home and during a diagnostic polysomnography in hospital. | 8 nights (7 nights at home and 1 night in the hospital)
  Comparison of the different oxygen parameters evaluated during 7 nights at home and during 1 night in the hospital
Variability in surrogate AHI | 7 nights
  Based on a previously developed algorithm, based on oximetry (including PPG), a surrogate AHI can be calculated. The variability in the surrogate AHI during 7 nights is evaluated.
Variability in cardiovascular comorbidity | 7 nights
  Based on a previously developed algorithm, based on oximetry (including PPG), the cardiovascular comorbidity can be estimated. The variability in this algorithm during 7 nights is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Bertien Buyse, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium